CLINICAL TRIAL: NCT00582192
Title: Seeking Informed Consent to Phase I Cancer Clinical Trials: Identifying Oncologists' Communication Styles
Brief Title: Seeking Informed Consent to Phase I Cancer Clinical Trials: Identifying Oncologists'Communication Styles
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Brown, Richard, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 07-096
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Cancer
Keywords: Phase I trial; Oncologists' Communication Styles
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Participants with certain types of cancers that are eligible for studies at Memorial Sloan-Kettering Cancer Center.
  Interventions: Other: Consult visit

INTERVENTIONS:
Other: Consult visit — Your appointment with your doctor will be audio taped. The research team will listen to the tape(s) and type them up. The team will then look for patterns in the discussions between patients and doctors. They will use this information to see if the discussions can be improved.

SUMMARY:
The purpose of this study is to examine doctor-patient communication about treatment options which may include an experimental, new treatment for cancer. What we learn from this study may help us to teach doctors better ways to talk to their patients.

DETAILED DESCRIPTION:
Subjects will be cancer patients attending one of three outpatient clinics at Memorial Sloan-Kettering Cancer Center. Subjects will be recruited from the Melanoma/Sarcoma, GI and Genitourinary Oncology services. The patients of six oncologists across the three services will be approached. All patients of these six oncologists who are invited to participate in a Phase I clinical trial will be approached to participate in the study. Patients who consent to participate in this study will be included in the sample regardless of their trial decision.

Design and Analysis:

To gather information about the communication strategies used by oncologists to discuss trials, a qualitative analysis of audio recordings of consultations containing discussions of Phase I trials will be conducted. These consultations will be audio recorded and transcribed in full; analysis will proceed using the constant comparative method. Initially (and as is consistent with the qualitative method employed for this study), a small sample of 15 patients will be recruited. Once an exhaustive analysis of this original data set is complete a further set of 15 patients will be recruited and transcripts of these consultations analyzed. In order to identify any new themes, the themes that emerged from the new data set will be compared with those identified in the original data set. We anticipate that the study will be completed within one year of commencement.

Significance: Oncologists report that one of their most significant communication challenges is communicating effectively and ethically with their patients about joining a clinical trial. Communication skills training has demonstrated efficacy in assisting doctors in this difficult task, however, there is a paucity of research in this area and studies have been limited to the Phase II and III trial setting. There is some research evidence that suggests that different communication issues and challenges emerge in the Phase I versus the Phase II and III trial setting. The pilot research proposed in this protocol will: a) explore the types of communication currently used by oncologists when recruiting patients to clinical trials and b) develop a set of communication strategies that can be used to address gaps in doctor- patient communication in this difficult area.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the outpatient oncology clinics of the six participating physicians (Drs Schwartz, Scher, Slovin, Tse, Shah & Carvajal)
* Diagnosed with cancer
* Eligible for a Phase I trial
* Discussing participation in such a trial with their physician during their visit

Exclusion Criteria:

* Fewer than 18 years of age
* Not proficient in English
* Cognitively or physically impaired, rendering them incapable of providing informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with certain types of cancers that are eligible for studies at Memorial Sloan-Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
This study aims to use qualitative research methods to examine the pattern of communication strategies oncologists use to discuss Phase I clinical trials ith their patients. | This study will begin with your appointment with your doctor the day of registration and will end at the end of the visit that day.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org